CLINICAL TRIAL: NCT05044104
Title: A Prospective Study of the Role and Accuracy of Consumer-Facing Wearable Technology in Gastrointestinal Endoscopy
Brief Title: Wearable Technology in Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Vinay Chandrasekhara, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-007738
Record Dates: First submitted 2021-09-04; First posted 2021-09-14 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Healthy
Keywords: Gastrointestinal Endoscopic Procedure with sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Wearable technology in endoscopic gastrointestinal procedures with sedation (Experimental): Subjects undergoing a endoscopic gastrointestinal procedure with sedation as part of standard of care will wear a consumer-facing wearable smart watch for the duration of the procedure.
  Interventions: Device: Consumer-facing wearable smart watch

INTERVENTIONS:
Device: Consumer-facing wearable smart watch — Wearable watch technology that has the ability to measure heart rate, respiratory rate, single-lead electrocardiography, and blood oxygen saturation.
  Other Names: Apple Watch Series 6; FitBit Versa

SUMMARY:
Researchers are assessing the accuracy and safety of wearable technology in subjects undergoing endoscopic gastrointestinal procedures with sedation.

DETAILED DESCRIPTION:
This is a prospective, non-blinded, exploratory study to assess the accuracy and safety of wearable devices in the endoscopy suite with patients undergoing procedures using anesthesia assisted sedation using smart watches. We will also simultaneously perform an assessment of patient and provider preferences using narrative-driven, qualitative evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years of age.
* Undergoing anesthesia-assisted endoscopic procedures.
* Able to give appropriate consent to the study or have an appropriate representative to do so.

Exclusion Criteria:

* Pregnancy.
* Physical deformity, wound, or dressing preventing placement of a wearable device on the wrist.
* Allergy to aluminum, nickel or acrylate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Chandrasekhara, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Undergoing Gastrointestinal Endoscopy With Sedation: Patients who underwent an endoscopic gastrointestinal procedure with sedation as part of standard of care who wore a consumer-facing wearable smart watch for the duration of the procedure.
Period: Overall Study
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Started | 292
Completed | 292
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Number analyzed (Participants) | 292
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.0 [45.8 to 71.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 173
  Male | 119
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Recorded Tachycardia Events
Description: Number of tachycardia events recorded as defined as heart rate > 100 bpm
Time Frame: Anesthesia Duration, approximately 30 to 45 minutes
Measure: Number; unit: Events
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Number analyzed (Participants) | 292
Events
  Anesthesia Monitoring | 9
  Smartwatch | 3
  Smartwatch Accessories | 22

2. Primary Outcome: Recorded Bradycardia Events
Description: Number of bradycardia events recorded as defined as heart rate < 60 bpm
Time Frame: Anesthesia Duration, approximately 30 to 45 minutes
Measure: Number; unit: Events
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Number analyzed (Participants) | 292
Events
  Anesthesia Monitoring | 119
  Smartwatch | 67
  Accessories | 33

3. Primary Outcome: Recorded Desaturation Events
Description: Number of desaturation events recorded as defined as peripheral O2 saturation <88%
Time Frame: Anesthesia Duration, approximately 30 to 45 minutes
Measure: Number; unit: events
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Number analyzed (Participants) | 292
events
  Anesthesia Monitoring | 91
  Smartwatch | 0
  Smartwatch Accessories | 71

4. Primary Outcome: Recorded Arrhythmia Events
Description: Number of arrhythmia events recorded
Time Frame: Anesthesia Duration, approximately 30 to 45 minutes
Measure: Number; unit: events
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Number analyzed (Participants) | 292
events
  Anesthesia Monitoring | 1
  Smartwatch | 0
  Smartwatch accessories | 0

5. Primary Outcome: Recorded Tachypnea
Description: Number of tachypnea events recorded as defined as respiratory rate >18 breaths per minute
Time Frame: Anesthesia Duration, approximately 30 to 45 minutes
Measure: Number; unit: events
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
Number analyzed (Participants) | 292
events
  Anesthesia Monitoring | 29
  Smartwatch | 0
  Smartwatch accessories | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study participation for a total of approximately 14 days on all participants.
Arm/Group | Patients Undergoing Gastrointestinal Endoscopy With Sedation
All-Cause Mortality (participants affected / at risk) | 0/292
Serious Adverse Events (participants affected / at risk) | 0/292
Other Adverse Events (participants affected / at risk) | 0/292

LIMITATIONS AND CAVEATS:
Limited number of arrhythmia events; Inconsistent accuracy of device reading; Device fit differed between patients

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-04): https://cdn.clinicaltrials.gov/large-docs/04/NCT05044104/Prot_SAP_000.pdf